#### **Original Article NCT03615755**

## Short Duration Hyperbaric Oxygen Therapy to Improve HbA1c, Leukocyte, and Serum Creatinine in Patient with Diabetic Foot Ulcer Wagner 3-4

#### **Author:**

#### dr. Hendry Irawan

Surgery Department, Faculty of Medicine, Udayana University, Sanglah General Hospital, Denpasar, Indonesia.

#### Co-Author 1:

#### Dr. dr. I Nyoman Semadi, Sp.B, Sp.BTKV

Thorax and Cardiovascular Surgery Division, Surgery Department, Faculty of Medicine, Udayana University, Sanglah General Hospital, Denpasar, Indonesia.

#### Co-Author 2:

#### Prof. Dr. dr. I Gde Raka Widiana, Sp.PD-KGH

Nephrology and Hypertension Division, Internal Medicine Department, Faculty of Medicine, Udayana University, Sanglah General Hospital, Denpasar, Indonesia.

#### **Correspondence:**

Name : dr. Hendry Irawan Phone : +62 82125097786

Email : <u>hendry irawan@rocketmail.com</u>

Affiliation : Surgery Department, Faculty of Medicine, Udayana University,

Sanglah General Hospital, Denpasar, Indonesia.

Address : Kesehatan Street No. 1, Denpasar, Bali, Indonesia.

Denpasar, 10-04-2018

dr. Hendry Irawan

#### **Results**

All patients were treated with insulin as antidiabetic and intravenous empiric antibiotics. We used combination short acting and long acting insulin daily. Dose of short acting (NovoRapid®, insulin aspart) 8 units every 8 hours and long acting (Lantus®, insulin glargine) 10 units at night. We grouped into two groups, each group consisted of 15 patients (**Table 1**), with mean age of standard therapy group  $56.67 \pm 8.30$  years old and combination therapy group  $50.53 \pm 7.52$  years old. Patients with the combination therapy group experienced longer DFUs  $6.07 \pm 4.13$  weeks than standard therapy group  $3.34 \pm 2.09$  weeks.

Analysis of HbA1c levels, leukocyte count, and serum creatinine levels were described in **Table 2**, **Table 3**, and **Table 4**. Comparison of baseline HbA1c levels between groups was not different with p = 0.059, but after two weeks there was significantly different between groups, p = 0.001 (**Table 2**). Evaluation pre and post therapy of HbA1c was significant in both of groups, in standard therapy group (from  $10.98 \pm 2.37$  % to  $9.70 \pm 2.46$  %; p = 0.006) and in combination therapy group (from  $9.42 \pm 1.96$  % to  $7.07 \pm 1.16$  %; p < 0.001).

Baseline of leukocyte count and the end of therapy between groups (**Table 3**) were not significant (p = 0.772 and p = 0.178, respectively), although leukocyte count after two weeks in combination therapy group decreased higher than standard therapy group. Leukocyte count in combination therapy group was significantly decreased from  $13.97 \pm 6.24 \times 10^3$  cells/ $\mu$ L to 8.84  $\pm$  2.88 x  $10^3$  cells/ $\mu$ L; p = 0.009. In this study, the effect size of HbA1c and leukocyte count was not significant difference. At the end of therapy, leukocyte count between debridement and debridement with amputation was not significant difference. In combination therapy, patients who did debridement had leukocyte count 8.63  $\pm$  3.04 x  $10^3$  cells/ $\mu$ L compared with debridement with toe amputation  $9.17 \pm 2.84 \times 10^3$  cells/ $\mu$ L. Compared with standard therapy, the leukocyte count was higher in debridement and debridement with amputation (11.2  $\pm$  6.30 x  $10^3$  cells/ $\mu$ L,  $10.74 \pm 4.62 \times 10^3$  cells/ $\mu$ L, respectively).

In **Table 4**, the baseline and after two weeks of serum creatinine levels were not comparable because in standard therapy group had good renal function, whereas in combination

therapy group had impaired renal function. In standard therapy group, serum creatinine levels were stable, but serum creatinine levels were little decreased in combination therapy group. The effect size was not significant decrease in serum creatinine level (p = 0.732) between groups.

Table 1. Characteristics of Patients

| | Standard therapy | Standard therapy + HBOT |
|---|---|---|
| Variables | (n=15) | (n=15) |
| Age (years old) <sup>a</sup> | $56.67 \pm 8.30$ | $50.53 \pm 7.52$ |
| Duration of DFU (weeks) <sup>a</sup> | $3.34 \pm 2.09$ | $6.07 \pm 4.13$ |
| Duration of DM (years) <sup>b</sup> | 4 (1-10) | 3 (0.17-25) |
| Body mass index (kg/m <sup>2</sup> ) <sup>b</sup> | 22.04 | 22.04 |
| , , | (14.33-36.73) | (17.58-29.40) |
| Sex (%) | | |
| Male | 4 (26.7) | 8 (53.3) |
| Female | 11 (73.3) | 7 (46.7) |
| Smoking (%) | | |
| Yes | 1 (6.7) | 3 (20) |
| No | 14 (93.3) | 12 (80) |
| Hypertension (%) | | |
| Yes | 6 (40) | 6 (40) |
| No | 9 (60) | 9 (60) |
| Ulcer classification (%) | | |
| Wagner 3 | 8 (53.3) | 6 (40) |
| Wagner 4 | 7 (46.7) | 9 (60) |
| Surgery (%) | | |
| Debridement | 9 (60) | 9 (60) |
| Debridement with toe amputation | 6 (40) | 6 (40) |
| Hemoglobin (g/dL) <sup>a</sup> | | |
| Baseline | $10.47\pm1.72$ | $10.34 \pm 1.55$ |
| After 2 weeks | $9.45 \pm 1.46$ | $11.04 \pm 1.47$ |
| Albumin (g/dL) <sup>a</sup> | | |
| Baseline | $3.00 \pm 0.56$ | $3.08 \pm 0.78$ |
| After 2 weeks | $3.07 \pm 0.53$ | $3.59 \pm 0.76$ |

<sup>a</sup>mean ± standard deviation; <sup>b</sup>median (range)

Table 2. HbA1c levels between groups

| HbA1c (%) | Standard | 95% | 6 CI | Combination | 95% | 6 CI | n |
|---|---|---|---|---|---|---|---|
| 110A1C (70) | therapy | Lower | Upper | therapy | Lower | Upper | р |
| Baseline | $10.98 \pm 2.37$ | 9.67 | 12.30 | $9.42 \pm 1.96$ | 8.33 | 10.50 | 0.059 |
| After 2 weeks | $9.70 \pm 2.46$ | 8.34 | 11.06 | $7.07 \pm 1.16$ | 6.43 | 7.72 | $0.001^{*}$ |
| Effect size | $1.28 \pm 1.54$ | 0.43 | 2.13 | $2.34 \pm 1.57$ | 1.47 | 3.21 | 0.072 |
| p | 0.006* | | | < 0.001* | | | |

All values were mean  $\pm$  standard deviation; \*p value < 0.05

Table 3. Leukocyte count between groups

| Leukocyte | Standard | 95% | 6 CI | Combination | 95% | 6 CI | n |
|---|---|---|---|---|---|---|---|
| $(10^3 \text{ cells/}\mu\text{L})$ | therapy | Lower | Upper | therapy | Lower | Upper | р |
| Baseline | $14.27 \pm 6.79$ | 10.51 | 18.03 | $13.97 \pm 6.24$ | 10.51 | 17.43 | 0.772 |
| After 2 weeks | $11.01 \pm 5.51$ | 7.96 | 14.07 | $8.84 \pm 2.88$ | 7.26 | 10.43 | 0.178 |
| Effect size | $3.26\pm7.76$ | -1.04 | 7.56 | $5.13 \pm 6.72$ | 1.40 | 8.85 | 0.468 |
| p | 0.14 | | | $0.009^{*}$ | | | |

All values were mean  $\pm$  standard deviation; \*p value < 0.05

Table 4. Serum creatinine levels between groups

| Serum creatinine | Standard | | | Combination | 95% | 6 CI | |
|---|---|---|---|---|---|---|---|
| (mg/dL) | therapy | | | therapy | Lower Upper | | p |
| Baseline | $0.73 \pm 0.27$ | 0.58 | 0.89 | $2.10 \pm 2.88$ | 0.50 | 3.69 | |
| After 2 weeks | $0.73 \pm 0.27$ | 0.58 | 0.89 | $2.05 \pm 2.77$ | 0.52 | 3.59 | |
| Effect size | $0 \pm 0.13$ | -0.07 | 0.07 | $0.05\pm0.45$ | -0.21 | 0.29 | 0.732 |
| р | 0.985 | | | 0.551 | | | |

All values were mean  $\pm$  standard deviation

#### DATA 30 SAMPEL

| | No | Name | Age | Sex | НВОТ |
|----|----|------|-----|-----|---------|
| 1 | 4 | MS | 57 | F | Control |
| 2 | 5 | DMW | 67 | F | Control |
| 3 | 23 | INS | 55 | М | Control |
| 4 | 25 | KB | 53 | М | Control |
| 5 | 26 | IAN | 71 | F | Control |
| 6 | 28 | IKS | 63 | F | Control |
| 7 | 29 | LP | 51 | F | Control |
| 8 | 30 | NKR | 48 | F | Control |
| 9 | 33 | INS | 55 | M | Control |
| 10 | 38 | NNS | 59 | F | Control |
| 11 | 43 | NWM | 59 | F | Control |
| 12 | 45 | RA | 46 | F | Control |
| 13 | 20 | NKR | 62 | F | Control |
| 14 | 21 | NK | 40 | M | Control |
| 15 | 22 | NKS | 64 | F | Control |
| 16 | 1 | KSS | 49 | F | НВОТ |
| 17 | 2 | WRA | 55 | M | НВОТ |
| 18 | 3 | MP | 42 | F | НВОТ |
| 19 | 9 | NKK | 43 | F | НВОТ |
| 20 | 10 | KS | 50 | M | HBOT |
| 21 | 14 | KS | 46 | F | HBOT |
| 22 | 15 | WS | 55 | M | HBOT |
| 23 | 16 | IMS | 55 | M | HBOT |
| 24 | 17 | MS | 64 | F | HBOT |
| 25 | 18 | MGS | 49 | M | HBOT |
| 26 | 24 | MW | 54 | M | HBOT |
| 27 | 32 | INS | 55 | M | HBOT |
| 28 | 34 | WS | 50 | F | HBOT |
| 29 | 36 | FF | 33 | F | HBOT |
| 30 | 40 | IWS | 58 | M | HBOT |

| | Smoking | Hypertension | DurDM | DurUlcer | Wagner | Foot |
|----|---------|--------------|-------|----------|--------|-------|
| 1 | No | Yes | 6.00 | 4.00 | 4 | Right |
| 2 | No | Yes | 10.0 | 6.00 | 4 | Right |
| 3 | No | Yes | 7.00 | 1.00 | 3 | Left |
| 4 | Yes | No | 3.00 | 2.00 | 4 | Right |
| 5 | No | No | 4.00 | 1.00 | 4 | Right |
| 6 | No | No | 8.00 | 6.00 | 3 | Right |
| 7 | No | No | 1.00 | 3.00 | 4 | Right |
| 8 | No | No | 3.00 | 2.00 | 3 | Left |
| 9 | No | Yes | 7.00 | 4.00 | 3 | Right |
| 10 | No | Yes | 3.00 | 1.00 | 3 | Right |
| 11 | No | No | 3.00 | 4.00 | 3 | Left |
| 12 | No | Yes | 10.0 | 2.14 | 3 | Right |
| 13 | No | No | 2.00 | 2.00 | 4 | Left |
| 14 | No | No | 9.00 | 8.00 | 3 | Right |
| 15 | No | No | 1.00 | 4.00 | 4 | Left |
| 16 | No | No | 3.00 | 8.00 | 4 | Left |
| 17 | Yes | No | 10.0 | 4.00 | 4 | Right |
| 18 | No | No | .17 | 8.00 | 4 | Right |
| 19 | No | No | 3.00 | 3.00 | 3 | Right |
| 20 | No | No | 5.00 | 8.00 | 4 | Left |
| 21 | No | No | 1.00 | 4.00 | 4 | Right |
| 22 | No | Yes | 25.0 | 6.00 | 4 | Right |
| 23 | No | No | .17 | 8.00 | 3 | Right |
| 24 | No | No | 3.00 | 1.00 | 3 | Left |
| 25 | No | Yes | 9.00 | 6.00 | 3 | Right |
| 26 | Yes | Yes | 14.0 | 1.00 | 4 | Left |
| 27 | No | Yes | .50 | 2.00 | 4 | Right |
| 28 | No | No | 5.00 | 4.00 | 3 | Left |
| 29 | No | Yes | 5.00 | 16.0 | 3 | Left |
| 30 | Yes | Yes | 2.50 | 12.0 | 4 | Left |

| | Weight | Height | Surgery | HbA1c_A | Hb_A | Leukocyte_A |
|----|--------|--------|-------------|---------|-------|-------------|
| 1 | 60 | 156 | Debri+amput | 8.83 | 9.18 | 19.50 |
| 2 | 60 | 160 | Debri+amput | 6.49 | 10.90 | 11.00 |
| 3 | 65 | 167 | Debridem | 10.50 | 10.22 | 32.32 |
| 4 | 60 | 175 | Debridem | 11.40 | 11.05 | 19.78 |
| 5 | 45 | 150 | Debri+amput | 15.40 | 12.83 | 14.19 |
| 6 | 60 | 160 | Debridem | 9.00 | 11.24 | 15.94 |
| 7 | 47 | 158 | Debridem | 13.10 | 9.75 | 21.31 |
| 8 | 55 | 157 | Debridem | 9.60 | 10.14 | 13.07 |
| 9 | 60 | 167 | Debri+amput | 9.80 | 9.96 | 9.37 |
| 10 | 60 | 165 | Debridem | 14.10 | 11.70 | 13.13 |
| 11 | 51 | 155 | Debridem | 10.20 | 7.22 | 11.15 |
| 12 | 100 | 165 | Debridem | 12.60 | 14.44 | 7.67 |
| 13 | 56 | 154 | Debri+amput | 9.70 | 9.48 | 12.30 |
| 14 | 39 | 165 | Debridem | 10.30 | 8.60 | 7.13 |
| 15 | 41 | 147 | Debri+amput | 13.70 | 10.33 | 6.24 |
| 16 | 60 | 165 | Debridem | 13.67 | 10.40 | 11.91 |
| 17 | 60 | 168 | Debri+amput | 10.15 | 9.00 | 12.25 |
| 18 | 50 | 155 | Debri+amput | 7.99 | 7.38 | 7.86 |
| 19 | 70 | 155 | Debridem | 11.96 | 10.80 | 10.62 |
| 20 | 45 | 160 | Debri+amput | 10.45 | 9.90 | 7.20 |
| 21 | 48 | 150 | Debridem | 10.11 | 10.69 | 13.13 |
| 22 | 53 | 161 | Debridem | 8.77 | 11.30 | 13.90 |
| 23 | 74 | 165 | Debridem | 10.70 | 10.20 | 11.68 |
| 24 | 70 | 160 | Debridem | 9.51 | 11.30 | 18.82 |
| 25 | 82 | 167 | Debridem | 6.83 | 8.10 | 19.30 |
| 26 | 65 | 175 | Debri+amput | 8.60 | 10.44 | 8.76 |
| 27 | 70 | 175 | Debri+amput | 7.30 | 12.06 | 31.85 |
| 28 | 70 | 160 | Debridem | 9.70 | 10.37 | 11.14 |
| 29 | 75 | 165 | Debridem | 9.40 | 13.80 | 19.19 |
| 30 | 50 | 160 | Debri+amput | 6.10 | 9.43 | 11.96 |

| | BUN_A | Cr_A | Albumin_A | HbA1c_B | Hb_B | Leukocyte_B |
|----|-------|------|-----------|---------|-------|-------------|
| 1 | 10 | .68 | 2.41 | 5.57 | 8.52 | 10.07 |
| 2 | 14 | .90 | 3.20 | 7.24 | 8.33 | 19.96 |
| 3 | 24 | 1.27 | 3.23 | 10.30 | 6.58 | 9.88 |
| 4 | 11 | .68 | 2.59 | 12.00 | 8.85 | 27.23 |
| 5 | 16 | .33 | 3.27 | 13.00 | 9.32 | 7.96 |
| 6 | 27 | 1.00 | 2.50 | 7.30 | 11.45 | 12.64 |
| 7 | 6 | .61 | 2.57 | 11.50 | 8.73 | 9.90 |
| 8 | 15 | .44 | 3.16 | 10.10 | 9.36 | 10.67 |
| 9 | 16 | 1.13 | 3.55 | 8.70 | 11.09 | 9.82 |
| 10 | 23 | 1.06 | 2.05 | 15.00 | 8.88 | 6.64 |
| 11 | 16 | .66 | 2.92 | 8.00 | 9.27 | 7.21 |
| 12 | 20 | .56 | 4.17 | 10.10 | 12.10 | 9.23 |
| 13 | 9 | .52 | 2.74 | 9.00 | 8.09 | 7.70 |
| 14 | 13 | .63 | 2.84 | 7.90 | 10.53 | 7.40 |
| 15 | 17 | .53 | 3.77 | 9.80 | 10.68 | 8.91 |
| 16 | 68 | 2.62 | 3.02 | 8.26 | 11.60 | 5.62 |
| 17 | 8 | .78 | 3.28 | 6.63 | 11.47 | 13.47 |
| 18 | 8 | .41 | 2.84 | 5.40 | 10.50 | 7.11 |
| 19 | 6 | .72 | 2.89 | 7.37 | 10.60 | 12.44 |
| 20 | 9 | .50 | 5.47 | 9.46 | 11.60 | 6.35 |
| 21 | 5 | .43 | 3.45 | 8.57 | 13.70 | 6.73 |
| 22 | 31 | 2.48 | 2.61 | 6.27 | 8.30 | 14.25 |
| 23 | 14 | 1.10 | 2.30 | 7.29 | 11.10 | 7.41 |
| 24 | 20 | .88 | 3.18 | 7.04 | 12.60 | 5.78 |
| 25 | 75 | 5.30 | 2.30 | 5.80 | 9.50 | 8.28 |
| 26 | 25 | 2.32 | 2.95 | 6.80 | 10.09 | 7.48 |
| 27 | 15 | 1.25 | 2.54 | 7.20 | 12.09 | 8.83 |
| 28 | 11 | .51 | 2.82 | 5.90 | 10.72 | 6.96 |
| 29 | 21 | .76 | 3.83 | 8.20 | 12.76 | 10.18 |
| 30 | 50 | 11.3 | 2.70 | 5.90 | 8.96 | 11.78 |

| | BUN_B | Cr_B | Albumin_B | BMI | decreased_HbA1c |
|----|-------|------|-----------|-------|-----------------|
| 1 | 12 | .90 | 2.83 | 24.65 | 3.26 |
| 2 | 24 | .78 | 2.98 | 23.44 | 75 |
| 3 | 17 | 1.17 | 3.10 | 23.31 | .20 |
| 4 | 5 | .54 | 2.30 | 19.59 | 60 |
| 5 | 3 | .41 | 2.37 | 20.00 | 2.40 |
| 6 | 25 | .90 | 2.60 | 23.44 | 1.70 |
| 7 | 2 | .46 | 3.42 | 18.83 | 1.60 |
| 8 | 12 | .50 | 2.66 | 22.31 | 50 |
| 9 | 15 | 1.21 | 3.91 | 21.51 | 1.10 |
| 10 | 9 | 1.05 | 2.92 | 22.04 | 90 |
| 11 | 10 | .65 | 3.73 | 21.23 | 2.20 |
| 12 | 6 | .47 | 3.47 | 36.73 | 2.50 |
| 13 | 4 | .43 | 2.76 | 23.61 | .70 |
| 14 | 25 | .91 | 3.02 | 14.33 | 2.40 |
| 15 | 18 | .63 | 3.97 | 18.97 | 3.90 |
| 16 | 34 | 2.14 | 3.75 | 22.04 | 5.41 |
| 17 | 14 | .70 | 3.20 | 21.26 | 3.52 |
| 18 | 15 | .76 | 3.97 | 20.81 | 2.59 |
| 19 | 35 | 1.74 | 3.90 | 29.14 | 4.59 |
| 20 | 10 | .75 | 3.41 | 17.58 | .99 |
| 21 | 11 | .59 | 4.06 | 21.33 | 1.54 |
| 22 | 70 | 2.30 | 1.50 | 20.45 | 2.50 |
| 23 | 27 | 1.19 | 4.19 | 27.18 | 3.41 |
| 24 | 9 | .75 | 3.85 | 27.34 | 2.47 |
| 25 | 71 | 4.19 | 4.61 | 29.40 | 1.03 |
| 26 | 23 | 2.07 | 3.31 | 21.22 | 1.80 |
| 27 | 13 | 1.08 | 3.56 | 22.86 | .10 |
| 28 | 13 | .44 | 3.43 | 27.34 | 3.80 |
| 29 | 18 | .71 | 4.43 | 27.55 | 1.20 |
| 30 | 55 | 11.4 | 2.72 | 19.53 | .20 |

| | decreased_leuko | decreased_Cr | increased_Hb |
|----|-----------------|--------------|--------------|
| 1 | 9.43 | 22 | 66 |
| 2 | -8.96 | .12 | -2.57 |
| 3 | 22.44 | .10 | -3.64 |
| 4 | -7.45 | .14 | -2.20 |
| 5 | 6.23 | 08 | -3.51 |
| 6 | 3.30 | .10 | .21 |
| 7 | 11.41 | .15 | -1.02 |
| 8 | 2.40 | 06 | 78 |
| 9 | 45 | 08 | 1.13 |
| 10 | 6.49 | .01 | -2.82 |
| 11 | 3.94 | .01 | 2.05 |
| 12 | -1.56 | .09 | -2.34 |
| 13 | 4.60 | .09 | -1.39 |
| 14 | 27 | 28 | 1.93 |
| 15 | -2.67 | 10 | .35 |
| 16 | 6.29 | .48 | 1.20 |
| 17 | -1.22 | .08 | 2.47 |
| 18 | .75 | 35 | 3.12 |
| 19 | -1.82 | -1.02 | 20 |
| 20 | .85 | 25 | 1.70 |
| 21 | 6.40 | 16 | 3.01 |
| 22 | 35 | .18 | -3.00 |
| 23 | 4.27 | 09 | .90 |
| 24 | 13.04 | .13 | 1.30 |
| 25 | 11.02 | 1.11 | 1.40 |
| 26 | 1.28 | .25 | 35 |
| 27 | 23.02 | .17 | .03 |
| 28 | 4.18 | .07 | .35 |
| 29 | 9.01 | .05 | -1.04 |
| 30 | .18 | 03 | 47 |

| | increased_Alb |
|----|---------------|
| 1 | .42 |
| 2 | 22 |
| 3 | 13 |
| 4 | 29 |
| 5 | 90 |
| 6 | .10 |
| 7 | .85 |
| 8 | 50 |
| 9 | .36 |
| 10 | .87 |
| 11 | .81 |
| 12 | 70 |
| 13 | .02 |
| 14 | .18 |
| 15 | .20 |
| 16 | .73 |
| 17 | 08 |
| 18 | 1.13 |
| 19 | 1.01 |
| 20 | -2.06 |
| 21 | .61 |
| 22 | -1.11 |
| 23 | 1.89 |
| 24 | .67 |
| 25 | 2.31 |
| 26 | .36 |
| 27 | 1.02 |
| 28 | .61 |
| 29 | .60 |
| 30 | .02 |

#### STATISTIC ANALISIS

# Explore HBOT

#### **Case Processing Summary**

| | Case F | rocessing | Julillary | | | | |
|---|---|---|---|---|---|---|---|
| | | | | Cas | ses | | |
| | | Valid | | Missing | | То | tal |
| | НВОТ | N | Percent | N | Percent | N | Percent |
| Age | НВОТ | 15 | 100.0% | 0 | .0% | 15 | 100.0% |
| | Control | 15 | 100.0% | 0 | .0% | 15 | 100.0% |
| Duration DM (years) | HBOT | 15 | 100.0% | 0 | .0% | 15 | 100.0% |
| | Control | 15 | 100.0% | 0 | .0% | 15 | 100.0% |
| Duration DFU (weeks) | НВОТ | 15 | 100.0% | 0 | .0% | 15 | 100.0% |
| | Control | 15 | 100.0% | 0 | .0% | 15 | 100.0% |
| HbA1c (%) pre | НВОТ | 15 | 100.0% | 0 | .0% | 15 | 100.0% |
| | Control | 15 | 100.0% | 0 | .0% | 15 | 100.0% |
| Hb (g/dL) pre | HBOT | 15 | 100.0% | 0 | .0% | 15 | 100.0% |
| | Control | 15 | 100.0% | 0 | .0% | 15 | 100.0% |
| Leukocyte (cells/uL) | HBOT | 15 | 100.0% | 0 | .0% | 15 | 100.0% |
| pre | Control | 15 | 100.0% | 0 | .0% | 15 | 100.0% |
| Creatinine (mg/dL) pre | HBOT | 15 | 100.0% | 0 | .0% | 15 | 100.0% |
| | Control | 15 | 100.0% | 0 | .0% | 15 | 100.0% |
| Albumin (g/dL) pre | HBOT | 15 | 100.0% | 0 | .0% | 15 | 100.0% |
| | Control | 15 | 100.0% | 0 | .0% | 15 | 100.0% |
| HbA1c (%) post | HBOT | 15 | 100.0% | 0 | .0% | 15 | 100.0% |
| | Control | 15 | 100.0% | 0 | .0% | 15 | 100.0% |
| Hb (g/dL) post | HBOT | 15 | 100.0% | 0 | .0% | 15 | 100.0% |
| | Control | 15 | 100.0% | 0 | .0% | 15 | 100.0% |
| Leukocyte (cells/uL) | HBOT | 15 | 100.0% | 0 | .0% | 15 | 100.0% |
| post | Control | 15 | 100.0% | 0 | .0% | 15 | 100.0% |
| Creatinine (mg/dL) | HBOT | 15 | 100.0% | 0 | .0% | 15 | 100.0% |
| post | Control | 15 | 100.0% | 0 | .0% | 15 | 100.0% |
| Albumin (g/dL) post | НВОТ | 15 | 100.0% | 0 | .0% | 15 | 100.0% |
| | Control | 15 | 100.0% | 0 | .0% | 15 | 100.0% |
| ВМІ | HBOT | 15 | 100.0% | 0 | .0% | 15 | 100.0% |
| | Control | 15 | 100.0% | 0 | .0% | 15 | 100.0% |

Descriptives<sup>a,b,c</sup>

| | НВОТ | | | Statistic | Std. Error |
|---|---|---|---|---|---|
| Age | НВОТ | <del>-</del> | Mean | 50.53 | 1.942 |
| | | 95% Confidence Interval for Mean | Lower Bound | 46.37 | |
| | | ioi ivicari | Upper Bound | 54.70 | |
| | | | 5% Trimmed Mean | 50.76 | |
| | | | Median | 50.00 | |
| | | | Variance | 56.552 | |

| | | _ | Std. Deviation | 7.520 | I |
|---|---|---|---|---|---|
| | | | Minimum | 33 | |
| | | | Maximum | 64 | |
| | | | Range | 31 | |
| | | | Interquartile Range | 9 | |
| | | | Skewness<br>Kurtosis | 636<br>1.082 | .580<br>1.121 |
| | Control | | Mean | 56.67 | 2.142 |
| | | 95% Confidence Interval | Lower Bound | 52.07 | |
| | | for Mean | Upper Bound | 61.26 | |
| | | | 5% Trimmed Mean | 56.80 | |
| | | | Median | 57.00 | |
| | | | Variance | 68.810 | |
| | | | Std. Deviation | 8.295 | |
| | | | Minimum | 40 | |
| | | | | l l | |
| | | | Maximum | 71 | |
| | | | Range | 31 | |
| | | | Interquartile Range | 12 | |
| | | | Skewness | 269 | .580 |
| Duration DM (years) | HBOT | <u> </u> | Kurtosis<br>Mean | 150<br>5.7560 | 1.121<br>1.71073 |
| | | 95% Confidence Interval | Lower Bound | 2.0869 | |
| | | for Mean | Upper Bound | 9.4251 | |
| | | | 5% Trimmed Mean | 4.9972 | |
| | | | Median | 3.0000 | |
| | | | Variance | 43.899 | |
| | | | Std. Deviation | 6.62563 | |
| | | | Minimum | .17 | |
| | | | Maximum | 25.00 | |
| | | | Range | 24.83 | |
| | | | Interquartile Range | 8.00 | |
| | | | Skewness | 2.011 | .580 |
| | | | Kurtosis | 4.540 | 1.121 |
| | Control | | Mean | 5.1333 | .82154 |
| | | 95% Confidence Interval for Mean | Lower Bound | 3.3713 | |
| | | | Upper Bound | 6.8954 | |
| | | | 5% Trimmed Mean | 5.0926 | |
| | | | Median | 4.0000 | |

| | | _ | | | |
|---|---|---|---|---|---|
| | | | Std. Deviation | 3.18179 | |
| | | | Minimum | 1.00 | |
| | | | Maximum | 10.00 | |
| | | | Range | 9.00 | |
| | | | Interquartile Range | 5.00 | |
| | | | Skewness | .290 | .580 |
| | | | Kurtosis | -1.408 | 1.121 |
| Duration DFU (weeks) | НВОТ | | Mean | 6.0667 | 1.06667 |
| | for Mean | Lower Bound | 3.7789 | | |
| | | | Upper Bound | 8.3544 | |
| | | | 5% Trimmed Mean | 5.7963 | |
| | | | Median | 6.0000 | |
| | | | Variance | 17.067 | |
| | | | Std. Deviation | 4.13118 | |
| | | | Minimum | 1.00 | |
| | | | Maximum | 16.00 | |
| | | | Range | 15.00 | |
| | | | Interquartile Range | 5.00 | |
| | | | Skewness | .976 | .580 |
| | | | Kurtosis | 1.047 | 1.121 |
| | Control | | Mean | 3.3427 | .53886 |
| | | 95% Confidence Interval for Mean | Lower Bound | 2.1869 | |
| | | ioi inidan | Upper Bound | 4.4984 | |
| | | | 5% Trimmed Mean | 3.2141 | |
| | | | Median | 3.0000 | |
| | | | Variance | 4.356 | |
| | | | Std. Deviation | 2.08701 | |
| | | | Minimum | 1.00 | |
| | | | Maximum | 8.00 | |
| | | | Range | 7.00 | |
| | | | Interquartile Range | 2.00 | |
| | | | Skewness | .835 | .580 |
| | | | Kurtosis | .130 | 1.121 |
| HbA1c (%) pre | НВОТ | | Mean | 9.4160 | .50556 |
| | | 95% Confidence Interval for Mean | Lower Bound | 8.3317 | |
| | | .s. moun | Upper Bound | 10.5003 | |
| | | | 5% Trimmed Mean | 9.3639 | |
| | | | Median | 9.5100 | |
| | | | | 1 | |
| | | | Variance | 3.834 | |

| | | | Minimum | 6.10 | |
|---|---|---|---|---|---|
| | | | Maximum | 13.67 | |
| | | | Range | 7.57 | |
| | | | Interquartile Range | 2.46 | |
| | | | Skewness | .335 | .580 |
| | | | Kurtosis | .449 | 1.121 |
| | Control | | Mean | 10.9813 | .61297 |
| | | 95% Confidence Interval for Mean | Lower Bound | 9.6666 | |
| | | | Upper Bound | 12.2960 | |
| | | | 5% Trimmed Mean | 10.9854 | |
| | | | Median | 10.3000 | |
| | | | Variance | 5.636 | |
| | | | Std. Deviation | 2.37402 | |
| | | | Minimum | 6.49 | |
| | | | Maximum | 15.40 | |
| | | | Range | 8.91 | |
| | | | Interquartile Range | 3.50 | |
| | | | Skewness | .215 | .580 |
| | | | Kurtosis | 275 | 1.121 |
| Hb (g/dL) pre | НВОТ | • | Mean | 10.3447 | .40082 |
| | | 95% Confidence Interval for Mean | Lower Bound | 9.4850 | |
| | | ior weari | Upper Bound | 11.2043 | |
| | | | 5% Trimmed Mean | 10.3174 | |
| | | | Median | 10.4000 | |
| | | | Variance | 2.410 | |
| | | | Std. Deviation | 1.55236 | |
| | | | Minimum | 7.38 | |
| | | | Maximum | 13.80 | |
| | | | Range | 6.42 | |
| | | | Interquartile Range | 1.87 | |
| | | | Skewness | .166 | .580 |
| | | | Kurtosis | 1.143 | 1.121 |
| | Control | | Mean | 10.4693 | .44524 |
| | | 95% Confidence Interval for Mean | Lower Bound | 9.5144 | |
| | | ioi weari | Upper Bound | 11.4243 | |
| | | | 5% Trimmed Mean | 10.4293 | |
| | | | Median | 10.2200 | |
| | | | Variance | 2.974 | |
| | | | Std. Deviation | 1.72442 | |
| | | | Minimum | 7.22 | |
| 1 | | | _ | | |

| | | _ | | _ | |
|---|---|---|---|---|---|
| | | | Maximum | 14.44 | |
| | | | Range | 7.22 | |
| | | | Interquartile Range | 1.76 | |
| | | | Skewness | .544 | .580 |
| Landa and Andrew Hallahala | LIDOT | | Kurtosis | 1.328 | 1.121 |
| Leukocyte (cells/uL) pre | HBOT | | Mean | 13.9713 | 1.61188 |
| | | 95% Confidence Interval for Mean | Lower Bound | 10.5142 | |
| | | | Upper Bound | 17.4285 | |
| | | | 5% Trimmed Mean | 13.3543 | |
| | | | Median | 11.9600 | |
| | | | Variance | 38.972 | |
| | | | Std. Deviation | 6.24278 | |
| | | | Minimum | 7.20 | |
| | | | Maximum | 31.85 | |
| | | | Range | 24.65 | |
| | | | Interquartile Range | 8.20 | |
| | | | Skewness | 1.811 | .580 |
| | | | Kurtosis | 4.101 | 1.121 |
| | Control | | Mean | 14.2733 | 1.75384 |
| | | 95% Confidence Interval<br>for Mean | Lower Bound | 10.5117 | |
| | | | Upper Bound | 18.0349 | |
| | | | 5% Trimmed Mean | 13.7170 | |
| | | | Median | 13.0700 | |
| | | | Variance | 46.139 | |
| | | | Std. Deviation | 6.79259 | |
| | | | Minimum | 6.24 | |
| | | | Maximum | 32.32 | |
| | | | Range | 26.08 | |
| | | | Interquartile Range | 10.13 | |
| | | | Skewness | 1.361 | .580 |
| | | | Kurtosis | 2.408 | 1.121 |
| Creatinine (mg/dL) pre | НВОТ | | Mean | 2.0953 | .74329 |
| | | 95% Confidence Interval | Lower Bound | .5011 | |
| | | for Mean | Upper Bound | 3.6895 | |
| | | | 5% Trimmed Mean | 1.6737 | |
| | | | Median | .8800 | |
| | | | Variance | 8.287 | |
| | | | Std. Deviation | 2.87877 | |
| | | | Minimum | .41 | |
| | | | Maximum | 11.37 | |
| | | | _ | 11.07 | |

| | | | | | - |
|---|---|---|---|---|---|
| | | | Range | 10.96 | |
| | | | Interquartile Range | 1.97 | |
| | | | Skewness | 2.773 | .580 |
| | | | Kurtosis | 8.306 | 1.121 |
| | Control | | Mean | .7333 | .07083 |
| | | 95% Confidence Interval for Mean | Lower Bound | .5814 | |
| | | | Upper Bound | .8852 | |
| | | | 5% Trimmed Mean | .7259 | |
| | | | Median | .6600 | |
| | | | Variance | .075 | |
| | | | Std. Deviation | .27432 | |
| | | | Minimum | .33 | |
| | | | Maximum | 1.27 | |
| | | | Range | .94 | |
| | | | Interquartile Range | .47 | |
| | | | Skewness | .629 | .580 |
| | | | Kurtosis | 589 | 1.121 |
| Albumin (g/dL) pre | НВОТ | - | Mean | 3.0787 | .20139 |
| | | 95% Confidence Interval for Mean | Lower Bound | 2.6467 | |
| | | ioi wean | Upper Bound | 3.5106 | |
| | | | 5% Trimmed Mean | 2.9891 | |
| | | | Median | 2.8900 | |
| | | | Variance | .608 | |
| | | | Std. Deviation | .77997 | |
| | | | Minimum | 2.30 | |
| | | | Maximum | 5.47 | |
| | | | Range | 3.17 | |
| | | | Interquartile Range | .67 | |
| | | | Skewness | 2.234 | .580 |
| | | | Kurtosis | 6.308 | 1.121 |
| | Control | · | Mean | 2.9980 | .14489 |
| | | 95% Confidence Interval | Lower Bound | 2.6872 | |
| | | for Mean | Upper Bound | 3.3088 | |
| | | | 5% Trimmed Mean | 2.9856 | |
| | | | Median | 2.9200 | |
| | | | Variance | .315 | |
| | | | Std. Deviation | .56117 | |
| | | | Minimum | 2.05 | |
| | | | Maximum | 4.17 | |
| | | | Range | 2.12 | |
| | | | - Kange | 2.12 | |

| | <u></u> | | | |
|---|---|---|---|---|
| | | Interquartile Range | .70 | |
| | | Skewness | .437 | .580 |
| LIDOT | | Kurtosis | | 1.121 |
| НВОТ | | | | .29966 |
| | 95% Confidence Interval for Mean | | | |
| | | Upper Bound | 7.7154 | |
| | | 5% Trimmed Mean | 7.0330 | |
| | | Median | 7.0400 | |
| | | Variance | 1.347 | |
| | | Std. Deviation | 1.16058 | |
| | | Minimum | 5.40 | |
| | | Maximum | 9.46 | |
| | | Range | 4.06 | |
| | | Interquartile Range | 2.30 | |
| | | Skewness | .502 | .580 |
| | | Kurtosis | 389 | 1.121 |
| Control | | Mean | 9.7007 | .63504 |
| | 95% Confidence Interval | Lower Bound | 8.3386 | |
| | ioi woan | Upper Bound | 11.0627 | |
| | | 5% Trimmed Mean | 9.6357 | |
| | | Median | 9.8000 | |
| | | Variance | 6.049 | |
| | | Std. Deviation | 2.45951 | |
| | | Minimum | 5.57 | |
| | | Maximum | 15.00 | |
| | | Range | 9.43 | |
| | | Interquartile Range | 3.60 | |
| | | Skewness | .508 | .580 |
| | | Kurtosis | .216 | 1.121 |
| НВОТ | | Mean | 11.0393 | .37848 |
| | 95% Confidence Interval | Lower Bound | 10.2276 | |
| | ioi wean | Upper Bound | 11.8511 | |
| | | 5% Trimmed Mean | 11.0437 | |
| | | Median | 11.1000 | |
| | | Variance | 2.149 | |
| | | Std. Deviation | 1.46584 | |
| | | Minimum | 8.30 | |
| | | Maximum | 13.70 | |
| | | Range | 5.40 | |
| | | Control 95% Confidence Interval for Mean Control 95% Confidence Interval for Mean | HBOT HBOT 95% Confidence Interval for Mean 95% Confidence Interval (Upper Bound 5% Trimmed Mean Median Variance Std. Deviation Minimum Maximum Range Interquartile Range Skewness Kurtosis Control 95% Confidence Interval for Mean 95% Confidence Interval for Mean Wedian Variance Std. Deviation Mean Upper Bound 5% Trimmed Mean Median Variance Std. Deviation Minimum Maximum Range Interquartile Range Skewness Kurtosis Mean P5% Confidence Interval For Mean Wedian Variance Std. Deviation Minimum Maximum Range Interquartile Range Skewness Kurtosis Mean P5% Confidence Interval For Mean P5% Confidence Interv | Skewness |

| | | _ | Skewness | 131 | .580 |
|---|---|---|---|---|---|
| | | | Kurtosis | 251 | 1.121 |
| | Control | | Mean | 9.4520 | .37707 |
| | | 95% Confidence Interval for Mean | Lower Bound | 8.6433 | |
| | | ioi ivieaii | Upper Bound | 10.2607 | |
| | | | 5% Trimmed Mean | 9.4644 | |
| | | | Median | 9.2700 | |
| | | | Variance | 2.133 | |
| | | | Std. Deviation | 1.46038 | |
| | | | Minimum | 6.58 | |
| | | | Maximum | 12.10 | |
| | | | Range | 5.52 | |
| | | | Interquartile Range | 2.16 | |
| | | | Skewness | .127 | .580 |
| | | | Kurtosis | 139 | 1.121 |
| Leukocyte (cells/uL) post | НВОТ | | Mean | 8.8447 | .74073 |
| | | for Mean | Lower Bound | 7.2560 | |
| | | | Upper Bound | 10.4334 | |
| | | | 5% Trimmed Mean | 8.7235 | |
| | | | Median | 7.4800 | |
| | | | Variance | 8.230 | |
| | | | Std. Deviation | 2.86884 | |
| | | | Minimum | 5.62 | |
| | | | Maximum | 14.25 | |
| | | | Range | 8.63 | |
| | | | Interquartile Range | 5.05 | |
| | | | Skewness | .789 | .580 |
| | | | Kurtosis | 784 | 1.121 |
| | Control | | Mean | 11.0147 | 1.42290 |
| | | 95% Confidence Interval for Mean | Lower Bound | 7.9628 | |
| | | | Upper Bound | 14.0665 | |
| | | | 5% Trimmed Mean | 10.3569 | |
| | | | Median | 9.8200 | |
| | | | Variance | 30.370 | |
| | | | Std. Deviation | 5.51088 | |
| | | | Minimum | 6.64 | |
| | | | Maximum | 27.23 | |
| | | | Range | 20.59 | |
| | | | Interquartile Range | 2.97 | |
| | | | Skewness | 2.321 | .580 |

| | | | Kurtosis | 5.350 | 1.121 |
|---|---|---|---|---|---|
| Creatinine (mg/dL) post | НВОТ | • | Mean | 2.0540 | .71459 |
| | | 95% Confidence Interval for Mean | Lower Bound | .5213 | |
| | | ioi Mean | Upper Bound | 3.5867 | |
| | | | 5% Trimmed Mean | 1.6244 | |
| | | | Median | 1.0800 | |
| | | | Variance | 7.660 | |
| | | | Std. Deviation | 2.76761 | |
| | | | Minimum | .44 | |
| | | | Maximum | 11.40 | |
| | | | Range | 10.96 | |
| | | | Interquartile Range | 1.43 | |
| | | | Skewness | 3.132 | .580 |
| | | | Kurtosis | 10.613 | 1.121 |
| | Control | · | Mean | .7340 | .07095 |
| | | 95% Confidence Interval for Mean | Lower Bound | .5818 | |
| | | ioi mean | Upper Bound | .8862 | |
| | | | 5% Trimmed Mean | .7256 | |
| | | | Median | .6500 | |
| | | | Variance | .076 | |
| | | | Std. Deviation | .27479 | |
| | | | Minimum | .41 | |
| | | | Maximum | 1.21 | |
| | | | Range | .80 | |
| | | | Interquartile Range | .44 | |
| | | | Skewness | .453 | .580 |
| | | | Kurtosis | -1.176 | 1.121 |
| Albumin (g/dL) post | НВОТ | | Mean | 3.5927 | .19609 |
| | | 95% Confidence Interval for Mean | Lower Bound | 3.1721 | |
| | | ioi modii | Upper Bound | 4.0132 | |
| | | | 5% Trimmed Mean | 3.6524 | |
| | | | Median | 3.7500 | |
| | | | Variance | .577 | |
| | | | Std. Deviation | .75946 | |
| | | | Minimum | 1.50 | |
| | | | Maximum | 4.61 | |
| | | | Range | 3.11 | |
| | | | Interquartile Range | .75 | |
| | | | Skewness | -1.480 | .580 |
| | | | Kurtosis | 3.353 | 1.121 |

| | Control | | Mean | 3.0693 | .13616 |
|---|---|---|---|---|---|
| | | 95% Confidence Interval | Lower Bound | 2.7773 | |
| | | for Mean | Upper Bound | 3.3614 | |
| | | | 5% Trimmed Mean | 3.0620 | |
| | | | Median | 2.9800 | |
| | | | Variance | .278 | |
| | | | Std. Deviation | .52734 | |
| | | | Minimum | 2.30 | |
| | | | Maximum | 3.97 | |
| | | | Range | 1.67 | |
| | | | Interquartile Range | .81 | |
| | | | Skewness | .396 | .580 |
| | | | Kurtosis | 831 | 1.121 |
| ВМІ | НВОТ | | Mean | 23.6690 | 1.00114 |
| | | 95% Confidence Interval for Mean | Lower Bound | 21.5218 | |
| | | ioi ivieari | Upper Bound | 25.8162 | |
| | | | 5% Trimmed Mean | 23.6889 | |
| | | | Median | 22.0386 | |
| | | | Variance | 15.034 | |
| | | | Std. Deviation | 3.87738 | |
| | | | Minimum | 17.58 | |
| | | | Maximum | 29.40 | |
| | | | Range | 11.82 | |
| | | | Interquartile Range | 6.53 | |
| | | | Skewness | .216 | .580 |
| | | | Kurtosis | -1.500 | 1.121 |
| | Control | | Mean | 22.2661 | 1.23499 |
| | | 95% Confidence Interval for Mean | Lower Bound | 19.6173 | |
| | | | Upper Bound | 24.9149 | |
| | | | 5% Trimmed Mean | 21.9037 | |
| | | | Median | 22.0386 | |
| | | | Variance | 22.878 | |
| | | | Std. Deviation | 4.78308 | |
| | | | Minimum | 14.33 | |
| | | | Maximum | 36.73 | |
| | | | Range | 22.41 | |
| | | | Interquartile Range | 3.85 | |
| | | | Skewness | 1.836 | .580 |
| | | Tooto of Normality b.c.d | Kurtosis | 6.336 | 1.121 |

| | | Kolmo | Kolmogorov-Smirnov <sup>a</sup> | | S | hapiro-Wil | k |
|---|---|---|---|---|---|---|---|
| | НВОТ | Statistic | df | Sig. | Statistic | df | Sig. |
| Age | НВОТ | .153 | 15 | .200* | .952 | 15 | .555 |
| | Control | .087 | 15 | .200* | .991 | 15 | 1.000 |
| Duration DM (years) | HBOT | .279 | 15 | .003 | .776 | 15 | .002 |
| | Control | .215 | 15 | .059 | .904 | 15 | .110 |
| Duration DFU (weeks) | НВОТ | .187 | 15 | .169 | .914 | 15 | .157 |
| | Control | .184 | 15 | .181 | .900 | 15 | .095 |
| HbA1c (%) pre | HBOT | .123 | 15 | .200* | .978 | 15 | .955 |
| | Control | .180 | 15 | .200* | .961 | 15 | .707 |
| Hb (g/dL) pre | HBOT | .136 | 15 | .200* | .966 | 15 | .794 |
| | Control | .132 | 15 | .200* | .966 | 15 | .803 |
| Leukocyte (cells/uL) | НВОТ | .238 | 15 | .022 | .819 | 15 | .006 |
| pre | Control | .172 | 15 | .200* | .893 | 15 | .074 |
| BUN (mg/dL) pre | HBOT | .227 | 15 | .036 | .790 | 15 | .003 |
| | Control | .155 | 15 | .200* | .971 | 15 | .870 |
| Creatinine (mg/dL) pre | HBOT | .294 | 15 | .001 | .612 | 15 | .000 |
| | Control | .244 | 15 | .017 | .929 | 15 | .268 |
| Albumin (g/dL) pre | HBOT | .198 | 15 | .117 | .781 | 15 | .002 |
| | Control | .114 | 15 | .200* | .977 | 15 | .949 |
| HbA1c (%) post | HBOT | .132 | 15 | .200* | .959 | 15 | .668 |
| | Control | .137 | 15 | .200* | .976 | 15 | .935 |
| Hb (g/dL) post | HBOT | .090 | 15 | .200* | .989 | 15 | .999 |
| | Control | .192 | 15 | .143 | .961 | 15 | .703 |
| Leukocyte (cells/uL) | HBOT | .216 | 15 | .058 | .882 | 15 | .050 |
| post | Control | .325 | 15 | .000 | .687 | 15 | .000 |
| Creatinine (mg/dL) | НВОТ | .331 | 15 | .000 | .565 | 15 | .000 |
| post | Control | .160 | 15 | .200 <sup>*</sup> | .906 | 15 | .119 |
| Albumin (g/dL) post | НВОТ | .169 | 15 | .200* | .893 | 15 | .073 |
| | Control | .143 | 15 | .200* | .948 | 15 | .487 |
| ВМІ | НВОТ | .217 | 15 | .055 | .889 | 15 | .065 |
| | Control | .256 | 15 | .009 | .802 | 15 | .004 |

a. Lilliefors Significance Correction

#### **Crosstabs**

#### **Case Processing Summary**

| | | | = | = | | |
|---------------------|----|---------|-----|---------|----|---------|
| | | Cases | | | | |
| | Va | lid | Mis | sing | To | tal |
| | N | Percent | N | Percent | N | Percent |
| SEX * HBOT | 30 | 100.0% | 0 | .0% | 30 | 100.0% |
| Smoking * HBOT | 30 | 100.0% | 0 | .0% | 30 | 100.0% |
| Hypertension * HBOT | 30 | 100.0% | 0 | .0% | 30 | 100.0% |
| Wagner * HBOT | 30 | 100.0% | 0 | .0% | 30 | 100.0% |

<sup>\*.</sup> This is a lower bound of the true significance.

#### **SEX \* HBOT**

#### Crosstab

| | _ | _ | HB | ОТ | |
|-----|--------|---------------|--------|---------|--------|
| | | | НВОТ | Control | Total |
| SEX | Male | Count | 8 | 4 | 12 |
| | | % within HBOT | 53.3% | 26.7% | 40.0% |
| | Female | Count | 7 | 11 | 18 |
| | | % within HBOT | 46.7% | 73.3% | 60.0% |
| · | Total | Count | 15 | 15 | 30 |
| | | % within HBOT | 100.0% | 100.0% | 100.0% |

## Smoking \* HBOT

#### Crosstab

| Ī | _ | - | НВ | НВОТ | |
|---------|-------|---------------|--------|---------|--------|
| | | | НВОТ | Control | Total |
| Smoking | Yes | Count | 3 | 1 | 4 |
| | | % within HBOT | 20.0% | 6.7% | 13.3% |
| | No | Count | 12 | 14 | 26 |
| | | % within HBOT | 80.0% | 93.3% | 86.7% |
| | Total | Count | 15 | 15 | 30 |
| | | % within HBOT | 100.0% | 100.0% | 100.0% |

## Hypertension \* HBOT

#### Crosstab

| | | | НВ | НВОТ | |
|--------------|-------|---------------|--------|---------|--------|
| | | | НВОТ | Control | Total |
| Hypertension | Yes | Count | 6 | 6 | 12 |
| | | % within HBOT | 40.0% | 40.0% | 40.0% |
| | No | Count | 9 | 9 | 18 |
| | | % within HBOT | 60.0% | 60.0% | 60.0% |
| | Total | Count | 15 | 15 | 30 |
| | | % within HBOT | 100.0% | 100.0% | 100.0% |

## Wagner \* HBOT

#### Crosstab

| | | | НВ | НВОТ | |
|--------|-------|---------------|--------|---------|--------|
| · | | | НВОТ | Control | Total |
| Wagner | 3 | Count | 6 | 8 | 14 |
| | | % within HBOT | 40.0% | 53.3% | 46.7% |
| | 4 | Count | 9 | 7 | 16 |
| | | % within HBOT | 60.0% | 46.7% | 53.3% |
| | Total | Count | 15 | 15 | 30 |
| | | % within HBOT | 100.0% | 100.0% | 100.0% |

## GROUP 1 (HBOT)

#### T-Test

#### **Paired Samples Statistics**

| | - | Mean | N | Std. Deviation | Std. Error Mean |
|--------|----------------|--------|----|----------------|-----------------|
| Pair 1 | HbA1c (%) pre | 9.4160 | 15 | 1.95802 | .50556 |
| | HbA1c (%) post | 7.0727 | 15 | 1.16058 | .29966 |

Paired Samples Test

| | | Paired Differences | | |
|---|---|---|---|---|
| | | Mean | Std. Deviation | Std. Error Mean |
| Pair 1 | HbA1c (%) pre - HbA1c (%)<br>post | 2.34333 | 1.57272 | .40607 |

#### **Paired Samples Test**

| | | Paired Differences | |
|---|---|---|---|
| | | 95% Confidence Interval of the<br>Difference | |
| | | Lower | Upper |
| Pair 1 | HbA1c (%) pre - HbA1c (%)<br>post | 1.47239 | 3.21427 |

**Paired Samples Test** 

| | | t | df | Sig. (2-tailed) |
|--------|-----------------------------------|-------|----|-----------------|
| Pair 1 | HbA1c (%) pre - HbA1c (%)<br>post | 5.771 | 14 | .000 |

#### **NPar Tests**

#### **Descriptive Statistics**

| | N | Mean | Std. Deviation | Minimum | Maximum |
|---|---|---|---|---|---|
| Leukocyte (cells/uL) pre | 15 | 13.9713 | 6.24278 | 7.20 | 31.85 |
| Creatinine (mg/dL) pre | 15 | 2.0953 | 2.87877 | .41 | 11.37 |
| Leukocyte (cells/uL) post | 15 | 8.8447 | 2.86884 | 5.62 | 14.25 |
| Creatinine (mg/dL) post | 15 | 2.0540 | 2.76761 | .44 | 11.40 |

#### Ranks

| | - | N | Mean Rank | Sum of Ranks |
|---|---|---|---|---|
| Leukocyte (cells/uL) post - | Negative Ranks | 12 <sup>d</sup> | 8.83 | 106.00 |
| Leukocyte (cells/uL) pre | Positive Ranks | 3 <sup>e</sup> | 4.67 | 14.00 |
| | Ties | Of | | |
| | Total | 15 | | |
| Creatinine (mg/dL) post - | Negative Ranks | 9 <sup>j</sup> | 7.83 | 70.50 |
| Creatinine (mg/dL) pre | Positive Ranks | 6 <sup>k</sup> | 8.25 | 49.50 |
| | Ties | OI | u<br>L | |
| | Total | 15 | | |

#### **Descriptive Statistics**

| | N | Mean | Std. Deviation | Minimum | Maximum |
|---|---|---|---|---|---|
| Leukocyte (cells/uL) pre | 15 | 13.9713 | 6.24278 | 7.20 | 31.85 |
| Creatinine (mg/dL) pre | 15 | 2.0953 | 2.87877 | .41 | 11.37 |
| Leukocyte (cells/uL) post | 15 | 8.8447 | 2.86884 | 5.62 | 14.25 |
| Creatinine (mg/dL) post | 15 | 2.0540 | 2.76761 | .44 | 11.40 |

#### Ranks

| | | N | Mean Rank | Sum of Ranks |
|---|---|---|---|---|
| Leukocyte (cells/uL) post - | Negative Ranks | 12 <sup>d</sup> | 8.83 | 106.00 |
| Leukocyte (cells/uL) pre | Positive Ranks | 3 <sup>e</sup> | 4.67 | 14.00 |
| | Ties | O <sup>f</sup> | | |
| | Total | 15 | | |
| Creatinine (mg/dL) post - | Negative Ranks | 9 <sup>j</sup> | 7.83 | 70.50 |
| Creatinine (mg/dL) pre | Positive Ranks | 6 <sup>k</sup> | 8.25 | 49.50 |
| | Ties | Ol | | |
| | Total | 15 | | |

- d. Leukocyte (cells/uL) post < Leukocyte (cells/uL) pre e. Leukocyte (cells/uL) post > Leukocyte (cells/uL) pre f. Leukocyte (cells/uL) post = Leukocyte (cells/uL) pre j. Creatinine (mg/dL) post < Creatinine (mg/dL) pre k. Creatinine (mg/dL) post > Creatinine (mg/dL) pre

- I. Creatinine (mg/dL) post = Creatinine (mg/dL) pre

#### Test Statistics<sup>c</sup>

| | Leukocyte<br>(cells/uL) post -<br>Leukocyte<br>(cells/uL) pre | Creatinine<br>(mg/dL) post -<br>Creatinine<br>(mg/dL) pre |
|---|---|---|
| Z | -2.613ª | 596ª |
| Asymp. Sig. (2-tailed) | .009 | .551 |

- a. Based on positive ranks.
- b. Based on negative ranks.
- c. Wilcoxon Signed Ranks Test

#### GROUP 2 (Control / Non HBOT)

#### T-Test

#### **Paired Samples Statistics**

| - | - | Mean | N | Std. Deviation | Std. Error Mean |
|---|---|---|---|---|---|
| Pair 1 | HbA1c (%) pre | 10.9813 | 15 | 2.37402 | .61297 |
| | HbA1c (%) post | 9.7007 | 15 | 2.45951 | .63504 |
| Pair 2 | Creatinine (mg/dL) pre | .7333 | 15 | .27432 | .07083 |
| | Creatinine (mg/dL) post | .7340 | 15 | .27479 | .07095 |

#### **Paired Samples Correlations**

| | - | N | Correlation | Sig. |
|---|---|---|---|---|
| Pair 1 | HbA1c (%) pre & HbA1c (%) post | 15 | .799 | .000 |
| Pair 2 | Creatinine (mg/dL) pre & Creatinine (mg/dL) post | 15 | .883 | .000 |

**Paired Samples Test** 

| | | Paired Differences | | |
|---|---|---|---|---|
| | | Mean | Std. Deviation | Std. Error Mean |
| Pair 1 | HbA1c (%) pre - HbA1c (%)<br>post | 1.28067 | 1.53573 | .39652 |
| Pair 2 | Creatinine (mg/dL) pre -<br>Creatinine (mg/dL) post | 00067 | .13258 | .03423 |

**Paired Samples Test** 

| | - | Paired Differences | |
|---|---|---|---|
| | | 95% Confidence Interval of th Difference Lower Upper | |
| Pair 1 | HbA1c (%) pre - HbA1c (%)<br>post | .43021 | 2.13113 |
| Pair 2 | Creatinine (mg/dL) pre -<br>Creatinine (mg/dL) post | 07409 | .07276 |

**Paired Samples Test** 

| | | t | df | Sig. (2-tailed) |
|---|---|---|---|---|
| Pair 1 | HbA1c (%) pre - HbA1c (%)<br>post | 3.230 | 14 | .006 |
| Pair 2 | Creatinine (mg/dL) pre -<br>Creatinine (mg/dL) post | 019 | 14 | .985 |

#### **NPar Tests**

#### **Descriptive Statistics**

| | N | Mean | Std. Deviation | Minimum | Maximum |
|---|---|---|---|---|---|
| Leukocyte (cells/uL) pre | 15 | 14.2733 | 6.79259 | 6.24 | 32.32 |
| Leukocyte (cells/uL) post | 15 | 11.0147 | 5.51088 | 6.64 | 27.23 |

## Wilcoxon Signed Ranks Test

#### Ranks

| | | N | Mean Rank | Sum of Ranks |
|---|---|---|---|---|
| Leukocyte (cells/uL) post - | Negative Ranks | 9 <sup>d</sup> | 9.56 | 86.00 |
| Leukocyte (cells/uL) pre | Positive Ranks | 6 <sup>e</sup> | 5.67 | 34.00 |
| | Ties | Of | | |
| | Total | 15 | | |

- d. Leukocyte (cells/uL) post < Leukocyte (cells/uL) pre
- e. Leukocyte (cells/uL) post > Leukocyte (cells/uL) pre
- f. Leukocyte (cells/uL) post = Leukocyte (cells/uL) pre

#### Test Statistics<sup>b</sup>

| | Leukocyte<br>(cells/uL) post -<br>Leukocyte<br>(cells/uL) pre |
|---|---|
| Z | -1.477ª |
| Asymp. Sig. (2-tailed) | .140 |

a. Based on positive ranks.

#### Ranks

| | | N | Mean Rank | Sum of Ranks |
|---|---|---|---|---|
| Leukocyte (cells/uL) post - | Negative Ranks | 9 <sub>q</sub> | 9.56 | 86.00 |
| Leukocyte (cells/uL) pre | Positive Ranks | 6e | 5.67 | 34.00 |
| | Ties | O <sup>f</sup> | | |
| | Total | 15 | | |

- d. Leukocyte (cells/uL) post < Leukocyte (cells/uL) pre
- e. Leukocyte (cells/uL) post > Leukocyte (cells/uL) pre
- b. Wilcoxon Signed Ranks Test

#### PRE POST TEST BETWEEN GROUPS

#### **T-Test**

#### **Group Statistics**

| | HBOT | N | Mean |
|----------------|---------|----|---------|
| HbA1c (%) pre | HBOT | 15 | 9.4160 |
| | Control | 15 | 10.9813 |
| HbA1c (%) post | НВОТ | 15 | 7.0727 |
| | Control | 15 | 9.7007 |

#### **Group Statistics**

| | НВОТ | Std. Deviation | Std. Error Mean |
|----------------|---------|----------------|-----------------|
| HbA1c (%) pre | НВОТ | 1.95802 | .50556 |
| | Control | 2.37402 | .61297 |
| HbA1c (%) post | НВОТ | 1.16058 | .29966 |
| | Control | 2.45951 | .63504 |

#### **Independent Samples Test**

| | | | | t-test for Equality of Means |
|---|---|---|---|---|
| | | F | Sig. | t |
| HbA1c (%) pre | Equal variances assumed | 1.002 | .325 | |
| | Equal variances not assumed | | | -1.970 |
| HbA1c (%) post | Equal variances assumed | 5.407 | .028 | -3.743 |
| | Equal variances not assumed | | | -3.743 |

#### **Independent Samples Test**

| | | t-test for Equality of Means | | |
|---|---|---|---|---|
| | | df Sig. (2-tailed) Mean Differe | | |
| HbA1c (%) pre | Equal variances assumed | 28 | .059 | -1.56533 |
| | Equal variances not assumed | 27.021 | .059 | -1.56533 |
| HbA1c (%) post | Equal variances assumed | 28 | .001 | -2.62800 |
| | Equal variances not assumed | 19.940 | .001 | -2.62800 |

#### **Independent Samples Test**

| | | | | e Interval of the<br>ence |
|---|---|---|---|---|
| | | Std. Error<br>Difference | Lower Upp | |
| HbA1c (%) pre | Equal variances assumed | .79456 | -3.19291 | .06224 |
| | Equal variances not assumed | .79456 | -3.19557 | .06490 |
| HbA1c (%) post | Equal variances assumed | .70219 | -4.06638 | -1.18962 |
| | Equal variances not assumed | .70219 | -4.09303 | -1.16297 |

#### NPar Tests

#### **Descriptive Statistics**

| | N | Mean | Std. Deviation | Minimum | Maximum |
|---|---|---|---|---|---|
| Leukocyte (cells/uL) pre | 30 | 14.1223 | 6.41186 | 6.24 | 32.32 |
| Creatinine (mg/dL) pre | 30 | 1.4143 | 2.12529 | .33 | 11.37 |
| Leukocyte (cells/uL) post | 30 | 9.9297 | 4.45560 | 5.62 | 27.23 |
| Creatinine (mg/dL) post | 30 | 1.3940 | 2.04569 | .41 | 11.40 |
| HBOT | 30 | 1.50 | .509 | 1 | 2 |

## Mann-Whitney Test

#### Ranks

| | НВОТ | N | Mean Rank | Sum of Ranks |
|---------------------------|---------|----|-----------|--------------|
| Leukocyte (cells/uL) pre | HBOT | 15 | 15.03 | 225.50 |
| | Control | 15 | 15.97 | 239.50 |
| | Total | 30 | | |
| Creatinine (mg/dL) pre | HBOT | 15 | 17.87 | 268.00 |
| | Control | 15 | 13.13 | 197.00 |
| | Total | 30 | | |
| Leukocyte (cells/uL) post | HBOT | 15 | 13.33 | 200.00 |
| | Control | 15 | 17.67 | 265.00 |
| | Total | 30 | | |
| Creatinine (mg/dL) post | HBOT | 15 | 19.00 | 285.00 |
| | Control | 15 | 12.00 | 180.00 |
| | Total | 30 | | |

#### Test Statistics<sup>b</sup>

| | Leukocyte<br>(cells/uL) pre | Creatinine<br>(mg/dL) pre | Leukocyte<br>(cells/uL) post | Creatinine<br>(mg/dL) post |
|---|---|---|---|---|
| Mann-Whitney U | 105.500 | 77.000 | 80.000 | 60.000 |
| Wilcoxon W | 225.500 | 197.000 | 200.000 | 180.000 |
| Z | 290 | -1.473 | -1.348 | -2.178 |
| Asymp. Sig. (2-tailed) | .772 | .141 | .178 | .029 |
| Exact Sig. [2*(1-tailed Sig.)] | .775ª | .148ª | .187ª | .029ª |

a. Not corrected for ties.

# Explore HBOT

#### **Case Processing Summary**

| | Ca | ses |
|------|-------|---------|
| НВОТ | Valid | Missing |

b. Grouping Variable: HBOT

| | | N | Percent | N | Percent |
|-----------------|---------|----|---------|---|---------|
| decreased_HbA1c | HBOT | 15 | 100.0% | 0 | .0% |
| | Control | 15 | 100.0% | 0 | .0% |
| decreased_leuko | HBOT | 15 | 100.0% | 0 | .0% |
| | Control | 15 | 100.0% | 0 | .0% |
| decreased_Cr | HBOT | 15 | 100.0% | 0 | .0% |
| | Control | 15 | 100.0% | 0 | .0% |

Case Processing Summary

| | - | Cases | | ses |
|-----------------|---------|-----------|----|---------|
| | | Total | | tal |
| | HBOT | N Percent | | Percent |
| decreased_HbA1c | HBOT | | 15 | 100.0% |
| | Control | | 15 | 100.0% |
| decreased_leuko | HBOT | | 15 | 100.0% |
| | Control | | 15 | 100.0% |
| decreased_Cr | HBOT | | 15 | 100.0% |
| | Control | | 15 | 100.0% |

Descriptives

| | Descriptives | | | |
|---|---|---|---|---|
| НВОТ | | | Statistic | Std. Error |
| decreased_HbA1c HBOT | | Mean | 2.3433 | .40607 |
| | 95% Confidence Interval | Lower Bound | 1.4724 | |
| | for Mean | Upper Bound | 3.2143 | |
| | | 5% Trimmed Mean | 2.2976 | |
| | | Median | 2.4700 | |
| | | Variance | 2.473 | |
| | | Std. Deviation | 1.57272 | |
| | | Minimum | .10 | |
| | | Maximum | 5.41 | |
| | | Range | 5.31 | |
| | Interquartile Range | 2.49 | | |
| | | Skewness | .383 | .580 |
| <u> </u> | | Kurtosis | 597 | 1.121 |
| Control | • | Mean | 1.2807 | .39652 |
| | 95% Confidence Interval | Lower Bound | .4302 | |
| | for Mean | Upper Bound | 2.1311 | |
| | | 5% Trimmed Mean | 1.2563 | |
| | | Median | 1.6000 | |
| | | Variance | 2.358 | |
| | | Std. Deviation | 1.53573 | |
| | | Minimum | 90 | |
| | | _ | | • |

| | | <del>_</del> | Maximum | 3.90 | |
|---|---|---|---|---|---|
| | | | Range | 4.80 | |
| | | | Interquartile Range | 2.90 | |
| | | | Skewness | 029 | .580 |
| | | | Kurtosis | -1.158 | 1.121 |
| decreased_leuko | HBOT | | Mean | 5.1267 | 1.73542 |
| | | 95% Confidence Interval | Lower Bound | 1.4046 | |
| | | for Mean | Upper Bound | 8.8488 | |
| | | | 5% Trimmed Mean | 4.5185 | |
| | | | Median | 4.1800 | |
| | | | Variance | 45.175 | |
| | | | Std. Deviation | 6.72124 | |
| | | | Minimum | -1.82 | |
| | | | Maximum | 23.02 | |
| | | | Range | 24.84 | |
| | | | Interquartile Range | 8.83 | |
| | | | Skewness | 1.464 | .580 |
| | | | Kurtosis | 2.382 | 1.121 |
| | Control | • | Mean | 3.2587 | 2.00389 |
| | 95% Confidence Interval for Mean | Lower Bound | -1.0393 | | |
| | | U | Upper Bound | 7.5566 | |
| | | 5% Trimmed Mean | 2.8719 | | |
| | | | Median | 3.3000 | |
| | | | Variance | 60.234 | |
| | | | Std. Deviation | 7.76104 | |
| | | | Minimum | -8.96 | |
| | | | Maximum | 22.44 | |
| | | | Range | 31.40 | |
| | | | Interquartile Range | 8.05 | |
| | | | Skewness | .781 | .580 |
| | | | Kurtosis | 1.652 | 1.121 |
| decreased_Cr | НВОТ | • | Mean | .0413 | .11652 |
| | | 95% Confidence Interval | Lower Bound | 2086 | |
| | | for Mean | Upper Bound | .2913 | |
| | | | 5% Trimmed Mean | .0409 | |
| | | | Median | .0700 | |
| | | | Variance | .204 | |
| | | | Std. Deviation | .45130 | |
| | | | Minimum | -1.02 | |
| | | | <b>-</b> | l l | |

| | <del>-</del> | Maximum | 1.11 | |
|---------|-------------------------|---------------------|--------|--------|
| | | Range | 2.13 | |
| | | Interquartile Range | .34 | |
| | | Skewness | .026 | .580 |
| | | Kurtosis | 3.239 | 1.121 |
| Control | | Mean | 0007 | .03423 |
| | 95% Confidence Interval | Lower Bound | 0741 | |
| | for Mean | Upper Bound | .0728 | |
| | | 5% Trimmed Mean | .0065 | |
| | | Median | .0100 | |
| | | Variance | .018 | |
| | | Std. Deviation | .13258 | |
| | | Minimum | 28 | |
| | | Maximum | .15 | |
| | | Range | .43 | |
| | | Interquartile Range | .18 | |
| | | Skewness | 815 | .580 |
| | | Kurtosis | 195 | 1.121 |

**Tests of Normality** 

| | - | Kolmogorov-Smirnov <sup>a</sup> | | |
|-----------------|---------|---------------------------------|----|-------|
| | НВОТ | Statistic | df | Sig. |
| decreased_HbA1c | HBOT | .104 | 15 | .200* |
| | Control | .144 | 15 | .200* |
| decreased_leuko | HBOT | .183 | 15 | .188 |
| | Control | .139 | 15 | .200* |
| decreased_Cr | HBOT | .189 | 15 | .158 |
| | Control | .220 | 15 | .050 |

a. Lilliefors Significance Correction

#### **Tests of Normality**

| | - | Shapiro-Wilk | | |
|-----------------|---------|--------------|----|------|
| | НВОТ | Statistic | df | Sig. |
| decreased_HbA1c | HBOT | .964 | 15 | .758 |
| | Control | .940 | 15 | .386 |
| decreased_leuko | HBOT | .864 | 15 | .028 |
| | Control | .952 | 15 | .561 |
| decreased_Cr | HBOT | .910 | 15 | .134 |
| | Control | .899 | 15 | .091 |

<sup>\*.</sup> This is a lower bound of the true significance.

## T-Test

#### **Group Statistics**

| | HBOT | N | Mean |
|-----------------|---------|----|--------|
| decreased_HbA1c | HBOT | 15 | 2.3433 |
| | Control | 15 | 1.2807 |
| decreased_Cr | HBOT | 15 | .0413 |
| | Control | 15 | 0007 |

#### **Group Statistics**

| | HBOT | Std. Deviation | Std. Error Mean |
|-----------------|---------|----------------|-----------------|
| decreased_HbA1c | HBOT | 1.57272 | .40607 |
| | Control | 1.53573 | .39652 |
| decreased_Cr | HBOT | .45130 | .11652 |
| | Control | .13258 | .03423 |

#### Independent Samples Test

| | | Levene's Test for Equality o<br>Variances | | t-test for Equality of Means |
|---|---|---|---|---|
| | | F | Sig. | t |
| decreased_HbA1c | Equal variances assumed | .006 | .939 | 1.872 |
| | Equal variances not assumed | | | 1.872 |
| decreased_Cr | Equal variances assumed | 3.920 | .058 | .346 |
| | Equal variances not assumed | | | .346 |

#### Independent Samples Test

| | | t-test for Equality of Means | | |
|---|---|---|---|---|
| | | df | Sig. (2-tailed) | Mean Difference |
| decreased_HbA1c | Equal variances assumed | 28 | .072 | 1.06267 |
| | Equal variances not assumed | 27.984 | .072 | 1.06267 |
| decreased_Cr | Equal variances assumed | 28 | .732 | .04200 |
| | Equal variances not assumed | 16.399 | .734 | .04200 |

#### **Independent Samples Test**

| | - | t-test for Equality of Means | | |
|---|---|---|---|---|
| | | | | e Interval of the rence |
| | | Std. Error<br>Difference | Lower | Upper |
| decreased_HbA1c | Equal variances assumed | .56756 | 09993 | 2.22527 |
| | Equal variances not assumed | .56756 | 09996 | 2.22529 |
| decreased_Cr | Equal variances assumed | .12145 | 20678 | .29078 |
| | Equal variances not assumed | .12145 | 21495 | .29895 |

#### **NPar Tests**

#### **Descriptive Statistics**

| | N | Mean | Std. Deviation | Minimum | Maximum |
|-----------------|----|--------|----------------|---------|---------|
| decreased_leuko | 30 | 4.1927 | 7.19649 | -8.96 | 23.02 |
| HBOT | 30 | 1.50 | .509 | 1 | 2 |

## **Mann-Whitney Test**

#### Ranks

| | НВОТ | N | Mean Rank | Sum of Ranks |
|-----------------|---------|----|-----------|--------------|
| decreased_leuko | HBOT | 15 | 16.67 | 250.00 |
| | Control | 15 | 14.33 | 215.00 |
| | Total | 30 | | |

#### Test Statistics<sup>b</sup>

| | decreased_leuko |
|--------------------------------|-----------------|
| Mann-Whitney U | 95.000 |
| Wilcoxon W | 215.000 |
| z | 726 |
| Asymp. Sig. (2-tailed) | .468 |
| Exact Sig. [2*(1-tailed Sig.)] | .486ª |

a. Not corrected for ties.

b. Grouping Variable: HBOT